CLINICAL TRIAL: NCT02131454
Title: Impact of Inhalation Technique Training on the Course of Asthma and Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Efficacy of Inhalation Technique Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marta Dąbrowska, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUM-TI
Record Dates: First submitted 2014-05-03; First posted 2014-05-06 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: asthma and COPD treatment; inhalation techniques; training of inhalation
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and Inhalation technique training (Experimental): Training in technique of drug inhalation in asthma and COPD patients and education about the role of inhalation therapy in the course of the disease.
  Interventions: Other: Inhalation technique training
- Education (No Intervention): Basic education about asthma and COPD.

INTERVENTIONS:
Other: Inhalation technique training — Training in inhalation technique in asthmatics and COPD patients
  Arms: Education and Inhalation technique training

SUMMARY:
Pharmacologic treatment of asthma and COPD is based mainly on inhalations. The aim of the study is to determine if short training of inhalation technique in patients with obstructive diseases may influence the course of asthma and COPD.

DETAILED DESCRIPTION:
Both asthma and COPD are common medical problems. Pharmacologic treatment of asthma and COPD is based mainly on inhalations. The inhalation technique is the key factor for effective management of bronchial obstruction. At the same time, a significant proportion of patients with asthma or COPD do not use inhalers properly.

The aim of the study is:

* to analyze the frequency and type of common mistakes in inhalation technique and
* to determine the impact of short individual training of inhalation technique on the course of asthma and COPD.

Fifty patients with asthma and 50 patients with COPD treated in the out-patient clinic or in the Department of Internal Medicine, Pneumonology and Allergology will be enrolled to the study.

The stage of severity (COPD) and control of the disease (asthma), quality of life, proper inhaler intake will be assessed at the study onset and at a second visit after 6 months.

At the second visit all patients will get a short, individual information about the etiology, course and general treatment plan of asthma / COPD. Patients will be randomized into two groups:

A. group of patients trained in proper inhalation technique B. group of patients without inhalation technique training Control visits will be held 3 and 6 months after training.

ELIGIBILITY:
Inclusion criteria:

* age of 18 - 80 years
* asthma or COPD diagnosed at least 6 months before study enrollment
* everyday usage of at least one of the following: pressured meter dose inhaler (pMDI) or dry powdered inhaler (Aerolizer, Handihaler, Disc or Turbuhaler)
* no other comorbidities that could influence learning of inhalation technique (psychiatric or neurologic disorders)

Exclusion criteria:

* age less than 18 or above 80 years
* lack of informed consent
* asthma or COPD diagnosed less than 6 months prior to screening visit
* coexistence of respiratory diseases other than asthma or COPD
* irregular use (not every day) of at least one inhaled drug
* treatment with inhalers other than: pMDI, Disc, Turbuhaler, Handihaler or Aerolizer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Asthma or COPD exacerbations | 6 months
  The number and severity of asthma and COPD exacerbations.

SECONDARY OUTCOMES:
Quality of life. | baseline, 3 months, 6 months
  Change from baseline in quality of life questionnaires:
  for asthma patients - Asthma Quality of Life Questionnaire for COPD patients - Saint George's Respiratory Questionnaire

OTHER OUTCOMES:
Disease control. | baseline , 3 months , 6 months
  Change from baseline in Asthma Control Test (ACT) or COPD Assessment Test (CAT)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Background] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Background] Press VG, Arora VM, Shah LM, Lewis SL, Charbeneau J, Naureckas ET, Krishnan JA. Teaching the use of respiratory inhalers to hospitalized patients with asthma or COPD: a randomized trial. J Gen Intern Med. 2012 Oct;27(10):1317-25. doi: 10.1007/s11606-012-2090-9. Epub 2012 May 17. PMID 22592354
- [Background] Al-Showair RA, Tarsin WY, Assi KH, Pearson SB, Chrystyn H. Can all patients with COPD use the correct inhalation flow with all inhalers and does training help? Respir Med. 2007 Nov;101(11):2395-401. doi: 10.1016/j.rmed.2007.06.008. Epub 2007 Jul 12. PMID 17629471
- [Derived] Dabrowska M, Luczak-Wozniak K, Miszczuk M, Domagala I, Lubanski W, Leszczynski A, Maskey-Warzechowska M, Rubinsztajn R, Hermanowicz-Salamon J, Krenke R. Impact of a Single Session of Inhalation Technique Training on Inhalation Skills and the Course of Asthma and COPD. Respir Care. 2019 Oct;64(10):1250-1260. doi: 10.4187/respcare.06740. Epub 2019 Jun 18. PMID 31213572